CLINICAL TRIAL: NCT06266117
Title: Investigation of Factors Affecting Pain, Anxiety, and Comfort Levels in Patients Undergoing Coronary Angiography
Brief Title: Pain, Anxiety, and Comfort Levels in Coronary Angiography
Status: Not yet recruiting | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Sponsor
Other Study IDs: SBF-HMS-GES-03
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Pain; Anxiety; Nursing Caries
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study was designed as a descriptive study. The universe of the study is İzzet Baysal Training and Research Hospital; It consists of patients who underwent coronary angiography in the coronary intensive care unit.

DETAILED DESCRIPTION:
In the first part, the descriptive information of the patients will be used, and in the second part, "Perianesthesia Comfort Scale", "State/Trait Anxiety Scale" and "General Comfort Scale (GAS)" adapted into Turkish by Üstündağ and Aslan in 2010 will be used. Visual Pain Scale will be used for pain measurement.

It is planned that the data for the Perianesthesia Comfort Scale (PCI) will be collected in the patient's room on the first postoperative day, in approximately 15 minutes, by face-to-face interview method.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years Conscious patients

Exclusion Criteria:

* Patients undergoing intubation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing coronary angiography in the coronary intensive care unit
Sampling Method: Probability Sample
Enrollment: 216 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Pain level | on the 1st postoperative days
  Visual Pain Scale
Anxiety | on the 1st postoperative days
  State/Trait Anxiety Scale
Comfort | on the 1st postoperative days
  Perianesthesia Comfort Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Abant Izzet Baysal University Faculty of Health Science, Bolu, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soysal GE, Demir Erbas S. Factors influencing pain, anxiety, and comfort in patients undergoing coronary angiography: A prospective observational study. Saudi Med J. 2025 Jun;46(6):679-687. doi: 10.15537/smj.2025.46.6.20240158. PMID 40516941